CLINICAL TRIAL: NCT05287581
Title: A Progressive Home-based Exercise Intervention for Persons With Systemic Lupus Erythematosus
Brief Title: Motivating Individuals With Lupus to Exercise
Acronym: MOVES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Lupus Foundation of America (Other)
Responsible Party: Principal Investigator, Dominique Kinnett-Hopkins, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HUM00207257
Record Dates: First submitted 2022-03-09; First posted 2022-03-18 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The experimental intervention is a 16-week progressive home-based exercise program in which participants are supported through seven coaching calls based on social cognitive theory and motivational interviewing principles. The individual sessions will provide tailored support for increasing physical activity behavior towards the recommended guidelines of at least 150 minutes of moderate aerobic activity and two strength-training sessions per week. There are no drugs involved in the intervention.
  Interventions: Behavioral: MOVES
- Waitlist Control (No Intervention): 24-week waitlist control condition

INTERVENTIONS:
Behavioral: MOVES — The experimental intervention is a 16-week progressive home-based exercise program in which participants are supported through seven coaching calls based on social cognitive theory and motivational interviewing principles. The individual sessions will provide tailored support for increasing physical activity behavior towards the recommended guidelines of at least 150 minutes of moderate aerobic activity and two strength-training sessions per week. There are no drugs involved in the intervention.
  Arms: Experimental

SUMMARY:
Physical activity and exercise are helpful for managing symptoms like fatigue in people living with systemic lupus erythematosus (lupus; SLE). Despite research supporting physical activity participation, people with lupus are often inactive and report being afraid to exercise. To that end, this project is a pilot randomized controlled trial for examining the efficacy of a home-based behavioral intervention based on social cognitive theory and motivational interviewing for increasing physical activity and decreasing fatigue.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Lupus
* be able to speak and read English
* being non-active defined as not engaging in regular activity (150 minutes or more of moderate physical activity per week)
* being impacted by fatigue defined as a score of 36 or higher on the fatigue severity scale

Exclusion Criteria:

* moderate or high risk for undertaking physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Change in physical activity over time | Baseline and 4 months
  Actigraph accelerometers will be worn by participants on an elastic belt around their waist for 7 days.
Change in Exercise over time | Baseline, 2, 4, and 6 months
  The Godin Leisure-Time Exercise Questionnaire (GLTEQ) will be administered. The GLTEQ measures the frequency of strenuous, moderate, and mild leisure activity performed for periods of 15 min or more over a usual week.

SECONDARY OUTCOMES:
Change in Fatigue Severity Scale over time | Baseline, 2, 4, and 6 months
  The Fatigue Severity Scale measures the severity of fatigue and its effect on a person's activity and lifestyle. The items are scored on a 7-point scale with 1 = strongly disagree and 7 = strongly agree.
  The minimum score is 9, and the maximum score possible is 63. The higher the score, the greater the fatigue severity

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No